CLINICAL TRIAL: NCT05432596
Title: A Phase 2b, Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Parallel-Group Study to Determine the Safety, Tolerability, Pharmacokinetics, and Efficacy of ATI-1777 in Patients 12 to 65 Years Old With Mild to Severe Atopic Dermatitis (AD)
Brief Title: Study of ATI-1777 in Patients 12 to 65 Years Old With Mild to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATI-1777-AD-202
Record Dates: First submitted 2022-06-01; First posted 2022-06-27 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Vehicle-controlled, Parallel-group Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ATI-1777 topical solution 2.0% w/w (BID) (Experimental): ATI-1777 topical solution 2.0% w/w, twice daily
  Interventions: Drug: ATI-1777 2.0% w/w
- ATI-1777 topical solution 1.0% w/w (BID) (Experimental): ATI-1777 topical solution 1.0% w/w, twice daily
  Interventions: Drug: ATI-1777 1.0% w/w
- ATI-1777 topical solution 0.5% w/w (BID) (Experimental): ATI-1777 topical solution 0.5% w/w, twice daily
  Interventions: Drug: ATI-1777 0.5% w/w
- Vehicle (BID) (Placebo Comparator): Vehicle topical solution, twice daily
  Interventions: Drug: Vehicle
- ATI-1777 topical solution 2.0% w/w (QD) (Experimental): ATI-1777 topical solution 2.0% w/w, once daily
  Interventions: Drug: ATI-1777 2.0% w/w
- Vehicle (QD) (Placebo Comparator): Vehicle topical solution, once daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: ATI-1777 2.0% w/w — ATI-1777 topical solution 2.0% w/w
  Arms: ATI-1777 topical solution 2.0% w/w (BID); ATI-1777 topical solution 2.0% w/w (QD)
Drug: ATI-1777 1.0% w/w — ATI-1777 topical solution 1.0% w/w
  Arms: ATI-1777 topical solution 1.0% w/w (BID)
Drug: ATI-1777 0.5% w/w — ATI-1777 topical solution 0.5% w/w
  Arms: ATI-1777 topical solution 0.5% w/w (BID)
Drug: Vehicle — Vehicle topical solution
  Arms: Vehicle (BID); Vehicle (QD)

SUMMARY:
This is a Phase 2b study to determine the safety, tolerability, pharmacokinetic (PK), and efficacy of ATI-1777 in patients 12 to 65 years old with mild to severe Atopic Dermatitis. Eligible participants will apply either ATI-1777 or Vehicle Topical Solution once daily or twice daily for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign the IRB approved ICF/assent prior to administration of study-related procedures.
2. Male patients or non-pregnant, non-nursing female patients 12 to 65 years old, inclusive, at the time of informed consent/assent.
3. Have at least a 6-month history of AD prior to the Screening Visit, and no significant AD flares for the 4 weeks prior to the Screening Visit.

Exclusion Criteria:

1. Unstable course of AD (spontaneously improving or rapidly deteriorating) based on the patient history or as determined by the investigator during the Screening Period.
2. Concomitant skin disease or clinically infected AD or presence of other skin disease in the area to be dosed that may interfere with study assessments.
3. Female patients who are pregnant, nursing, or planning to become pregnant during the study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in Eczema Area and Severity Index Score (EASI) score at Week 4 (Day 28) | Baseline to Day 28
  EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD). The EASI score examines 4 areas of the body and weights them for participants 8 years of age and older as follows: Head/Neck (H) = 0.1, Upper limbs (UL) = 0.2, Trunk (T) = 0.3, and Lower limbs (LL) = 0.4. The severity strata for the EASI are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The total EASI score ranges from 0 to 72. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.

SECONDARY OUTCOMES:
Percentage change from baseline in EASI score at each post-baseline study visit | Baseline to Day 42
Proportion achieving Investigator's Global Assessment-Treatment Success (IGA-TS) defined as Validated Investigator Global Assessment (vIGA) score of 0 or 1 with an improvement in vIGA of at least 2 points from baseline at each post-baseline study visit. | Baseline to Day 42
  IGA is an assessment scale used to determine severity of atopic dermatitis (AD) and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). An IGA responder was defined as a participant achieving an IGA score of 0 to 1 and an IGA score improvement at least 2 from baseline.
Proportion of patients who achieve 50%, 75%, and 90% improvement in EASI score (EASI 50, EASI 75, and EASI 90, respectively) at each post-baseline study visit | Baseline to Day 42
Change from baseline in vIGA score at each post-baseline study visit | Baseline to Day 42
Change from baseline in Body Surface Area (BSA) at each post-baseline study visit | Baseline to Day 42
  BSA is defined as a percentage of the total body (0-100) that is affected by disease
Number of Participants With At Least One Adverse Event (AEs) and as Per Severity | Baseline to Day 42
  AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent. The severity of AEs was assessed using CTCAE v4.03 Grades 1 through 4.Data are reported for Grade 3 and higher severity for this outcome measure.
Change from baseline in Itch Numerical Rating Scale (PP NRS) from baseline to Day 28 | Baseline to Day 28
  The Itch NRS is a once-per-24 hours ("daily") participant-reported measure of itch intensity to rate the itching severity because of their AD by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best describes their worst level of itching in the past 24 hours. The categorical NRS is defined as 0 = None, 1 to 3 = Mild, 4 to 6 = Moderate, and 7 to 10 = Severe.study visit

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Aclaris Investigational Site, Birmingham, Alabama
  - Aclaris Investigational Site, Scottsdale, Arizona
  - Aclaris Investigational Site, Bryant, Arkansas
  - Aclaris Investigational Site, North Little Rock, Arkansas
  - Aclaris Investigational Site, Encinitas, California
  - Aclaris Investigational Site, Encino, California
  - Aclaris Investigational Site, Castle Rock, Colorado
  - Aclaris Investigational Site, Colorado Springs, Colorado
  - Aclaris Investigational Site, Delray Beach, Florida
  - Aclaris Investigational Site, Miami, Florida
  - Aclaris Investigational Site, Miami Lakes, Florida
  - Aclaris Investigational Site, Tampa, Florida
  - Aclaris Investigational Site, West Palm Beach, Florida
  - Aclaris Investigational Site, Sandy Springs, Georgia
  - Aclaris Investigational Site, Normal, Illinois
  - Aclaris Investigational Site, Skokie, Illinois
  - Aclaris Investigational Site, Indianapolis, Indiana
  - Aclaris Investigational Site, New Albany, Indiana
  - Aclaris Investigational Site, West Lafayette, Indiana
  - Aclaris Investigational Site, Baton Rouge, Louisiana
  - Aclaris Investigational Site, Houma, Louisiana
  - Aclaris Investigational Site, Saint Joseph, Missouri
  - Aclaris Investigational Site, Wilmington, North Carolina
  - Aclaris Investigational Site, Oklahoma City, Oklahoma
  - Aclaris Investigational Site, Medford, Oregon
  - Aclaris Investigational Site, Greenville, South Carolina
  - Aclaris Investigational Site, Murfreesboro, Tennessee
  - Aclaris Investigational Site, Arlington, Texas
  - Aclaris Investigational Site, Dallas, Texas
  - Aclaris Investigational Site, Houston, Texas
  - Aclaris Investigational Site, San Antonio, Texas
  - Aclaris Investigational Site, Richmond, Virginia